CLINICAL TRIAL: NCT06054828
Title: Modified Hospital Elder Life Program at Intensive Care Unit: A Stepped-Wedge Cluster Randomized Controlled Trial
Brief Title: Modified Hospital Elder Life Program at Intensive Care Unit
Acronym: mHelp@ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202301153RINB
Record Dates: First submitted 2023-08-08; First posted 2023-09-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: ICU Delirium
Keywords: Delirium; Intensive care units; Intervention; Mortality; Mobility; Cognitive function; Stepped-wedge cluster randomized controlled trial
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHELP@ICU (Experimental): Participants will receive cognitive engagement twice daily, have physical activity once daily, and be monitored for their feeding. The intervention will be administered for 14 days or until hospital discharge or death.
  Interventions: Behavioral: mHELP@ICU
- Control group (No Intervention): Participants in the control group will receive the usual care.

INTERVENTIONS:
Behavioral: mHELP@ICU — The 14-day mHELP@ICU consists of the following three components:
  1. Cognitive engagement twice daily: Participants will receive orienting communication, plus one of the following training on attention, memory, or function execution.
  2. Physical activity once daily: Participants will receive a passive range of motion(ROM) and/or anti-gravity ROM exercise if tolerated.
  3. Feeding monitor daily: The exact feeding data will be abstracted from medical records.
  Arms: mHELP@ICU

SUMMARY:
Delirium, a form of acute brain dysfunction, occurs in up to 81% of patients receiving mechanical ventilation in the intensive care unit (ICU). Delirium occurring in the ICU is associated with increased functional dependency, cognitive impairment, longer length of hospital stay, and mortality. This study aim to develop a nursing-driven ICU delirium intervention to reduce incidence of delirium, increase the delirium-and coma-free days (DCFDs), and improve ICU patients' function, cognition, and mortality outcomes 3 months following their ICU admission. The "modified Hospital Elder life Program at the ICU (mHELP@ICU)" will be provided to ensure critically ill patients are cognitively engaged, physically active, and nutritionally well-fed.

This three-year study is divided into two phases. The first phase aims to ensure the accuracy of delirium assessment using the Intensive Care Delirium Screening Checklist (ICDSC) by ICU nurses of three participating ICUs. The ICDSC records assessed by ICU nurses will be abstracted from medical records and compared with a gold standard ICDSC evaluation by a well-trained, independent assessor. Cohen's kappa will be reported to represent the consistency of the ICDSC assessment between delirium data from medical records and the independent assessor. When the Cohen's kappa is less than 0.8, a 3-month bedside teaching and real-time feedback education program will be implemented at three ICU units to improve the accuracy of ICDSC assessment by ICU nurses. The second phase will be a clinical trial using a stepped-wedge cluster randomized controlled trial design. Adult (18 years and older) critically ill patients receiving mechanical ventilation will be consecutively enrolled from three mix-medical ICUs at a studied medical center. Estimated 266 participants will be cluster-randomized into the intervention and control groups. Participants in the intervention group will receive a 14-day mHELP@ICU, provided by a trained mHELP nurse, while the participants who received the usual care will serve as controls. Effects of mHELP@ICU will be evaluated using the daily delirium and coma data (max 14 days, or until death or ICU discharge) retrieved from the medical records, along with the participants' mortality, cognitive, and functional outcomes, which a blinded outcome assessor will assess at 48 hours, 14 days, 30 days, and 90 days after ICU admission.

ELIGIBILITY:
Inclusion Criteria of the second phase

* participants who are 18 years old or older.
* participants who receive oral endotracheal intubation with mechanical ventilation and are expected intubation greater than 48 hours.
* participants are free from delirium or coma before ICU admission.

Exclusion Criteria of the second phase

* participants who are placed on droplet or contact precautions (e.g., Open TB, SARS, COVID-19 )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ICU delirium | Admitted to ICU for 14 days
  Delirium (yes/no) using ICDSC will be abstracted from medical records.
ICU delirium days | Admitted to ICU for 14 days
  Delirium (yes/no) using ICDSC will be abstracted from medical records.
Incidence of ICU coma | Admitted to ICU for 14 days
  Coma (yes/no) defined by RASS score of -4 or -5 will be abstracted from medical records.
ICU coma days | Admitted to ICU for 14 days
  Coma (yes/no) defined by RASS score of -4 or -5 will be abstracted from medical records.
Days of delirium- and coma-free days (DCFDs) | Admitted to ICU for 14 days
  DCFDs (yes/no) are defined as the number of days during the study period during which the patient was alive without delirium or coma associated with any cause and obtained.
Mortality | Admitted to ICU for 90 days
  Data will be obtained from medical records or participants' families.
Length of hospital stay | At hospital discharge
  Data will be obtained from medical records.

SECONDARY OUTCOMES:
Medical Research Council (MRC) score | At baseline (ICU admission); post-ICU 48 hours; day 30 and day 90 since ICU admission.
  Participants' muscle strength will be evaluated using the medical research council scale (MRC). Score range from 0 to 60; a higher score indicates better muscle strength.
Functional Status Score for the Intensive Care Unit (FSS-ICU) | At baseline (ICU admission); post-ICU 48 hours; day 30 and day 90 since ICU admission.
  Participants' functional status will be evaluated using the FSS-ICU. Score range from 0 to 35, a higher score indicates better functional status.
30-second sit-to-stand test | Post-ICU 48 hours; day 30 and day 90 since ICU admission.
  Participants will be asked for sit-to-stand repeatedly for 30 seconds.
Barthel index for activities of daily living (ADL) | At baseline (ICU admission); post-ICU 48 hours; day 30 and day 90 since ICU admission.
  Measured by ADL in score, range from 0-100 score, higher score indicated health condition
Montreal Cognitive Assessment (MoCA) | Post-ICU 48 hours; day 30 and day 90 since ICU admission.
  Participants' cognitive function will be evaluated using th MoCA. Score range from 0-30 score, higher than 23.5 scores indicates normal cognitive.
Color Trails Test (CTT) | Post-ICU 48 hours; day 30 and day 90 since ICU admission.
  Participants' visual attention and effortful executive processing abilities will be evaluated using the CTT; the time taken to complete each part of the CTT is recorded in seconds and is compared to normative data.
Accuracy rate of ICDSC data (yes/no) | Randomly select four days per week to verify the accuracy of ICDSC data during the first three months of the study.
  The ICDSC records assessed by ICU nurses will be abstracted from medical records and compared with a gold standard ICDSC evaluation by a well-trained, independent assessor.

CONTACTS AND LOCATIONS:
Locations (1):
- Cheryl, Chia-Hui Chen, PhD, Taipei, National Taiwan University, Taiwan

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Yamamoto T, Mizobata Y, Kawazoe Y, Miyamoto K, Ohta Y, Morimoto T, Yamamura H. Incidence, risk factors, and outcomes for sepsis-associated delirium in patients with mechanical ventilation: A sub-analysis of a multicenter randomized controlled trial. J Crit Care. 2020 Apr;56:140-144. doi: 10.1016/j.jcrc.2019.12.018. Epub 2019 Dec 24. PMID 31901649
- [Background] Fiest KM, Soo A, Hee Lee C, Niven DJ, Ely EW, Doig CJ, Stelfox HT. Long-Term Outcomes in ICU Patients with Delirium: A Population-based Cohort Study. Am J Respir Crit Care Med. 2021 Aug 15;204(4):412-420. doi: 10.1164/rccm.202002-0320OC. PMID 33823122
- [Background] Lat I, McMillian W, Taylor S, Janzen JM, Papadopoulos S, Korth L, Ehtisham A, Nold J, Agarwal S, Azocar R, Burke P. The impact of delirium on clinical outcomes in mechanically ventilated surgical and trauma patients. Crit Care Med. 2009 Jun;37(6):1898-905. doi: 10.1097/CCM.0b013e31819ffe38. PMID 19384221
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Brummel NE, Girard TD, Ely EW, Pandharipande PP, Morandi A, Hughes CG, Graves AJ, Shintani A, Murphy E, Work B, Pun BT, Boehm L, Gill TM, Dittus RS, Jackson JC. Feasibility and safety of early combined cognitive and physical therapy for critically ill medical and surgical patients: the Activity and Cognitive Therapy in ICU (ACT-ICU) trial. Intensive Care Med. 2014 Mar;40(3):370-9. doi: 10.1007/s00134-013-3136-0. Epub 2013 Nov 21. PMID 24257969
- [Background] Balas MC, Pun BT, Pasero C, Engel HJ, Perme C, Esbrook CL, Kelly T, Hargett KD, Posa PJ, Barr J, Devlin JW, Morse A, Barnes-Daly MA, Puntillo KA, Aldrich JM, Schweickert WD, Harmon L, Byrum DG, Carson SS, Ely EW, Stollings JL. Common Challenges to Effective ABCDEF Bundle Implementation: The ICU Liberation Campaign Experience. Crit Care Nurse. 2019 Feb;39(1):46-60. doi: 10.4037/ccn2019927. PMID 30710036
- [Background] Kotfis K, Marra A, Ely EW. ICU delirium - a diagnostic and therapeutic challenge in the intensive care unit. Anaesthesiol Intensive Ther. 2018;50(2):160-167. doi: 10.5603/AIT.a2018.0011. Epub 2018 Jun 8. PMID 29882581
- [Background] Maldonado JR. Delirium pathophysiology: An updated hypothesis of the etiology of acute brain failure. Int J Geriatr Psychiatry. 2018 Nov;33(11):1428-1457. doi: 10.1002/gps.4823. Epub 2017 Dec 26. PMID 29278283
- [Background] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Background] Hshieh TT, Yang T, Gartaganis SL, Yue J, Inouye SK. Hospital Elder Life Program: Systematic Review and Meta-analysis of Effectiveness. Am J Geriatr Psychiatry. 2018 Oct;26(10):1015-1033. doi: 10.1016/j.jagp.2018.06.007. Epub 2018 Jun 26. PMID 30076080
- [Background] American Geriatrics Society. AGS COCARE® . 2022
- [Background] Ely EW. The ABCDEF Bundle: Science and Philosophy of How ICU Liberation Serves Patients and Families. Crit Care Med. 2017 Feb;45(2):321-330. doi: 10.1097/CCM.0000000000002175. PMID 28098628
- [Background] Trogrlic Z, van der Jagt M, Bakker J, Balas MC, Ely EW, van der Voort PH, Ista E. A systematic review of implementation strategies for assessment, prevention, and management of ICU delirium and their effect on clinical outcomes. Crit Care. 2015 Apr 9;19(1):157. doi: 10.1186/s13054-015-0886-9. PMID 25888230
- [Background] Zhang S, Han Y, Xiao Q, Li H, Wu Y. Effectiveness of Bundle Interventions on ICU Delirium: A Meta-Analysis. Crit Care Med. 2021 Feb 1;49(2):335-346. doi: 10.1097/CCM.0000000000004773. PMID 33332818
- [Background] Chen CC, Li HC, Liang JT, Lai IR, Purnomo JDT, Yang YT, Lin BR, Huang J, Yang CY, Tien YW, Chen CN, Lin MT, Huang GH, Inouye SK. Effect of a Modified Hospital Elder Life Program on Delirium and Length of Hospital Stay in Patients Undergoing Abdominal Surgery: A Cluster Randomized Clinical Trial. JAMA Surg. 2017 Sep 1;152(9):827-834. doi: 10.1001/jamasurg.2017.1083. PMID 28538964
- [Background] Li HC, Yeh TY, Wei YC, Ku SC, Xu YJ, Chen CC, Inouye S, Boehm LM. Association of Incident Delirium With Short-term Mortality in Adults With Critical Illness Receiving Mechanical Ventilation. JAMA Netw Open. 2022 Oct 3;5(10):e2235339. doi: 10.1001/jamanetworkopen.2022.35339. PMID 36205994
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge trials using the Shiny CRT Calculator. Int J Epidemiol. 2020 Jun 1;49(3):979-995. doi: 10.1093/ije/dyz237. PMID 32087011
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Cowan SL, Preller J, Goudie RJB. Evaluation of the E-PRE-DELIRIC prediction model for ICU delirium: a retrospective validation in a UK general ICU. Crit Care. 2020 Mar 30;24(1):123. doi: 10.1186/s13054-020-2838-2. No abstract available. PMID 32228666
- [Background] Li HC, Chen CC, Yeh TY, Liao SC, Hsu AS, Wei YC, Shun SC, Ku SC, Inouye SK. Predicting hospital mortality and length of stay: A prospective cohort study comparing the Intensive Care Delirium Screening Checklist versus Confusion Assessment Method for the Intensive Care Unit. Aust Crit Care. 2023 May;36(3):378-384. doi: 10.1016/j.aucc.2022.01.010. Epub 2022 Mar 7. PMID 35272910
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Zaal IJ, Devlin JW, Peelen LM, Slooter AJ. A systematic review of risk factors for delirium in the ICU. Crit Care Med. 2015 Jan;43(1):40-7. doi: 10.1097/CCM.0000000000000625. PMID 25251759
- [Background] Park SY, Lee HB. Prevention and management of delirium in critically ill adult patients in the intensive care unit: a review based on the 2018 PADIS guidelines. Acute Crit Care. 2019 May;34(2):117-125. doi: 10.4266/acc.2019.00451. Epub 2019 Apr 17. PMID 31723916
- [Background] Abdulla H, Smith K, Atherton PJ, Idris I. Role of insulin in the regulation of human skeletal muscle protein synthesis and breakdown: a systematic review and meta-analysis. Diabetologia. 2016 Jan;59(1):44-55. doi: 10.1007/s00125-015-3751-0. Epub 2015 Sep 24. PMID 26404065
- [Background] De Jonghe B, Appere-De-Vechi C, Fournier M, Tran B, Merrer J, Melchior JC, Outin H. A prospective survey of nutritional support practices in intensive care unit patients: what is prescribed? What is delivered? Crit Care Med. 2001 Jan;29(1):8-12. doi: 10.1097/00003246-200101000-00002. PMID 11176150
- [Background] Uozumi M, Sanui M, Komuro T, Iizuka Y, Kamio T, Koyama H, Mouri H, Masuyama T, Ono K, Lefor AK. Interruption of enteral nutrition in the intensive care unit: a single-center survey. J Intensive Care. 2017 Aug 4;5:52. doi: 10.1186/s40560-017-0245-9. eCollection 2017. PMID 28794882
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Stollings JL, Kotfis K, Chanques G, Pun BT, Pandharipande PP, Ely EW. Delirium in critical illness: clinical manifestations, outcomes, and management. Intensive Care Med. 2021 Oct;47(10):1089-1103. doi: 10.1007/s00134-021-06503-1. Epub 2021 Aug 16. PMID 34401939